CLINICAL TRIAL: NCT03212729
Title: Antimicrobial Photodynamic Therapy Associated With the Conventional Endodontic Treatment: A Clinical and Molecular Microbiological Study
Brief Title: Antimicrobial Photodynamic Therapy Associated With the Conventional Endodontic Treatment: A Clinical and Microbiological Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Natalia Iorio Lopes Pontes Póvoa, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aPDT and microorganisms
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Photochemotherapy Reaction; Dental Pulp Necrosis; Polymerase Chain Reaction; Infection; Enterococcal Infections; Candida
MeSH Terms: conditions — Dental Pulp Necrosis; Infections; Torulopsis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): CONVENTIONAL ENDODONTIC TREATMENT
  Interventions: Procedure: Conventional endodontic treatment
- Test Group (Experimental): CONVENTIONAL ENDODONTIC TREATMENT ASSOCIATED WITH ANTIMICROBIAL PHOTODYNAMIC THERAPY
  Interventions: Radiation: ANTIMICROBIAL PHOTODYNAMIC THERAPY; Procedure: Conventional endodontic treatment

INTERVENTIONS:
Radiation: ANTIMICROBIAL PHOTODYNAMIC THERAPY — The aPDT was performed with 0.01% methylene blue and irradiated with low-level laser therapy (InGaAIP, 660 nm; 100 mW; 40 sec) with an optical fiber-coupled. Another irradiation (3 J; 30 sec; spot size of 3 mm2) was performed in the gingiva close to the apical foramen.
  Arms: Test Group
Procedure: Conventional endodontic treatment — After local anesthesia the supragingival calculus, biofilm and the carious tissues were removed. The access cavity preparation was completed. The crown-down technique was performed using Gates Glidden and Kerr files with an anatomic diameter compatible to the radicular canal, and the irrigation was performed with 5 mL of 2.5% NaOCl solution between each endodontic file. The working length was established 1 mm short of the radiographic apex. Smear layer was removed by rinsing the canal with 17% ethylene diamine tetra-acetic acid solution, which was left in the canal for 5 min, followed by a final irrigation with 15 mL of 2.5% NaOCl solution. Calcium hydroxide paste with paramonoclorophenol, was inserted into the canal, filling the root canal as temporary medication between the sessions. The coronal sealing was performed using Coltosol, followed by glass ionomer Maxxion R. Seven days later the root canal was filled by the hybrid Tagger technique, with a Mc Spadden condenser.

SUMMARY:
Microorganisms play a critical role in the etiology and pathogenesis of apical periodontitis. Enterococcus faecalis and Candida sp. are frequently associated with persistent infections. The aim of this study was evaluated the antimicrobial photodynamic therapy (aPDT) as an adjunct of the endodontic treatment. Ten uniradicular teeth [control group (CG)=4 and test group (TG)=6] with primary endodontic infections were analyzed. Microbiological samples were collected before and after the chemical-mechanical instrumentation (CMI), after the aPDT (for the TG) and after the temporary restorations removal (second session).

ELIGIBILITY:
Inclusion Criteria:

* Patients with teeth with: single canal with endodontic infection, intact pulp chamber walls, necrotic pulp confirmed by sensitivity pulp tests, and clinical and radiographic evidence of asymptomatic apical periodontitis

Exclusion Criteria:

* Patients with teeth with: gross carious lesions, root or crown fracture, previous endodontic treatment, gingival recession and periodontal pockets deeper than 4 mm.
* Patients pregnant, lactating, with systemic diseases that could compromise the immune system, individuals who received antibiotic therapy within the previous 3 months or in immunosuppressive treatment.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Antimicrobial photodynamic therapy (aPDT) evaluation on microorganisms erradication in canal roots after endodontic tretament and immediately use aPDT | Microorganisms detection were evaluated one month later
  The presence or absence of E. faecalis, Candida spp. and bacteria domains in the microbiological samples was determined by using end-point PCR. Aliquots of 10 ng of the extracted DNA were used in PCR protocols for E. faecalis, Candida genus and microorganisms from bacterial domains. Positive controls consisted of DNA extracted from E. faecalis (ATCC 29212) for detection of E. faecalis species and domain bacteria and C. albicans (ATCC 10321) for Candida genus. PCR amplifications were performed in a DNA thermocycler. Amplified products were analyzed by 1% of agarose gel electrophoresis with GelRed 1X and visualized on a UV transilluminator.